CLINICAL TRIAL: NCT01700972
Title: Feasibility and Diagnostic Accuracy of Myocardial SPECT Using Early Imaging Protocol: A Pilot Study
Brief Title: Feasibility and Diagnostic Accuracy of Myocardial Perfusion Imaging Using Early Imaging Protocol
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study did not recruit/no study activity occurred.
Sponsor: St. Louis University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REGA-12B03
Record Dates: First submitted 2012-08-14; First posted 2012-10-04 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging at 10-minute vs. 30-45-minutes (Experimental): The radionuclide Myoview will be administered once for the rest and stress myocardial perfusion imaging. The subsequent rest and stress imaging will be performed twice each - at 10 minutes and 30-45 minutes after radiotracer injection.
  Interventions: Procedure: Myocardial perfusion imaging

INTERVENTIONS:
Procedure: Myocardial perfusion imaging — The radionuclide Myoview will be administered once for the rest and stress myocardial perfusion imaging. The subsequent rest and stress imaging will be performed twice each - at 10 minutes and 30-45 minutes after radiotracer injection.
  Other Names: Myocardial perfusion SPECT

SUMMARY:
The current protocol for myocardial perfusion imaging (MPI) entails imaging within 30-45 minutes after radiotracer injection, for both rest and stress studies. We hypothesize that early imaging 10 minutes after radiotracer injection provides high image quality and diagnostic accuracy comparable to 30-45 minutes MPI.

DETAILED DESCRIPTION:
The current MPI protocol entails imaging within 30-45 minutes after radiotracer injection (W30 imaging), for both the rest and stress part. This delay between the radiotracer injection and imaging is intended to limit the nonspecific liver and gut radioactivity to the heart and allows an optimal imaging of the heart. A recent publication however indicates that an early imaging within 10 minutes after radiotracer injection (W10 imaging) appears feasible and may be as good as W30 imaging.

Encouraged by the recent data, we think that a waiting time of 10 minutes is feasible while preserving the image quality; thus, we would like to assess the feasibility and accuracy of W10 imaging compared with W30 imaging in this study. The main purpose of this study is to obtain imaging information on the use of early imaging (W10). The feasibility of W10 imaging will be assessed visually using a 3-point scale as well as semiquantitatively using region-of-interest measurements. The accuracy of W10 imaging will be determined by comparing the findings of W10 with those of coronary angiography, which will be obtained within 30 days of the MPI and serve as reference standard. The tolerability of W10 will be assessed using 3-point scale Questionnaires.

This study will determine if early MPI imaging within 10 minutes works as well as imaging after 30-45 minutes waiting and its role in the diagnosis of coronary artery disease. The major advantages of this new imaging procedure include the shortening of the procedure time, the reduction of patient discomfort and improvement of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age of any race /ethnicity
* Patient has undergone or is being scheduled for a clinically indicated cardiac catheterization with or without angioplasty
* Patient may have suffered myocardial infarction more than 3 days before MPI
* Patient may have undergone percutaneous transluminal coronary angioplasty (PTCA) or coronary stent placement more than 3 days prior to MPI
* Interval between T99m-MPI and cardiac catheterization is within 30 days
* Females are not pregnant and lactating
* Provide signed Informed Consent prior to undergoing the study procedures

Exclusion Criteria:

* Patients less than 18 years of age
* Female patient is pregnant or nursing
* Patient has been involved in any other investigative, radioactive research procedure within 7 days and during the study participation period
* History of 2nd or 3rd degree AV-block, or sinus node dysfunction unless the patients have a functioning artificial pacemaker
* Myocardial infarction within 3 days before MPI
* Percutaneous transluminal coronary angioplasty (PTCA) or stent placement within 3 days prior to MPI
* Current ventricular tachycardia, atrial fibrillation, atrial tachycardia, or atrial flutter
* Current history of exacerbated COPD or asthma
* Known hypersensitivity or contraindication to regadenoson or aminophylline
* Use of caffeinated substance, dipyridamole-containing medication, aminophylline, or xanthines containing medication (e.g. theophylline) within the 12 hours prior to Lexiscan administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility and accuracy of early imaging at 10 minutes (W10) vs. standard imaging at 30-45 minute after radiotracer injection | 30 days
  The feasibility of W10 imaging will be assessed visually using a 3-point scale as well as semiquantitatively using region-of-interest measurements. The accuracy of W10 imaging will be determined by comparing the findings of W10 with those of coronary angiography, which will be obtained within 30 days of the MPI and serve as reference standard.

SECONDARY OUTCOMES:
Tolerability of early imaging at 10 minutes (W10) | Two hours
  The tolerability of W10 will be assessed using 3-point scale Questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Nghi Nguyen, MD, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University School of Medicine, St Louis, Missouri, United States